CLINICAL TRIAL: NCT02090946
Title: The Experiences of Parents Learning Physiotherapy Techniques for Their Child
Status: Completed | Type: Observational
Sponsor: Western Sussex Hospitals NHS Trust (Other)
Collaborators: Brighton & Sussex Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 1507/WSHT/2012 and 11/163/WIL
Record Dates: First submitted 2013-12-13; First posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Developmental Disabilities
Keywords: children with physical disabilities; home activity programs; home programmes; learning; therapeutic relationship; phenomenology; physiotherapy; clinicians who teach; parent perspective; parent-professional relationships; Parents/carers; long term physiotherapy needs
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- parental experiences: interviews

SUMMARY:
The experiences of learning from paediatric physiotherapists were explored through unstructured interviews applying Colazzi's method to interpret the data. In this hermeneutic phenomenological study, six parents responsible for a physiotherapy home programme for their child were selected through convenience sampling. The purpose of this study was to obtain rich and valid information that could be analysed. The phenomenon of their learning experiences was formed and explored, its implications discussed and inferences made in light of current physiotherapy service delivery.

ELIGIBILITY:
Inclusion Criteria:

* parent/main carer of a child with a long term physical condition receiving physiotherapy in the United Kingdom for at least six months.

Exclusion Criteria:

* parents experiencing physiotherapy outside UK practice.
* parents to whom English is not their first language.
* parents under 16 years of age

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: convenience sample from the Arun, Adur and Worthing region, UK.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
the learning experiences of parents | after six months of physiotherapy
  using Colazzi's analysis interviews are coded and relevant data formed into themes that form the phenomenon.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Wilson, Principal Investigator — Western Sussex Hospitals NHS Foundation Trust
Locations (1):
- Western Sussex Hospitals NHS Foundation Trust, Worthing, West Sussex, United Kingdom

REFERENCES:
- [Result] Wilson, D. The learning Experiences of Parents whose Children require Physiotherapy Intervention. The Association of Paediatric Chartered Physiotherapists Journal 4 (2): 68, Nov, 2013